CLINICAL TRIAL: NCT02820662
Title: Study of the Implication of Omega-3 Polyunsaturated Fatty Acids in Retinopathy of Prematurity in Newborns
Brief Title: Study of the Implication of Omega-3 Polyunsaturated Fatty Acids in Retinopathy of Prematurity in New-born Infants
Acronym: OMEGAROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KOEHRER APJ 2014
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Blood Specimen Collection

ARMS (1):
- RETCAM (Experimental)
  Interventions: Other: RETCAM; Biological: Blood samples

INTERVENTIONS:
Other: RETCAM
Biological: Blood samples

SUMMARY:
The development of the retinal vascular network is generally complete during the 3rd trimester of pregnancy but may continue during the first 15 days of life. This late maturation may cause problems in pre-term births and may result in immature vascularization of the retina, a condition called retinopathy of prematurity. Among the different factors affecting the development of the retinal vasculature, the tissue level of omega-3 polyunsaturated fatty acids (PUFA) appears to be a crucial element, as does the form of the PUFA present in the tissues (nature of the phospholipids in their membranes). This project aims to show a possible association between levels of omega-3 PUFA and the onset of retinopathy of prematurity (ROP).

ELIGIBILITY:
Inclusion Criteria:

* Premature new-born infants born at less than 29 weeks of amenorrhea after informed consent has been obtained from a parent or the legal guardian of the infant

Exclusion Criteria:

* Premature new-born infants presenting a life-threatening condition. Persons without national health insurance cover

Ages: 0 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Stage of retinopathy of prematurity using a Retcam according to the ICROP classification (International Classification of Retinopathy of Prematurity) revised in 2005. | At 4 weeks of life or 31 weeks of amenorrhea

SECONDARY OUTCOMES:
Concentrations of omega-3 PUFA in Red Blood Cell (RBC) membranes. | At inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France

REFERENCES:
- [Result] Pallot C, Soudry Faure A, Charvy C, Ternoy N, Langlet Muteau C, Acar N, Bron AM, Speeg Schatz C, Creuzot-Garcher C. Screening for Retinopathy of Prematurity: Insight into Optimizing Screening. Ophthalmic Res. 2018;59(4):228-234. doi: 10.1159/000477622. Epub 2017 Jul 27. PMID 28746942